CLINICAL TRIAL: NCT04992676
Title: Comorbid Insomnia and Sleep Disordered Breathing in Patients Undergoing Cardiac Rehabilitation: Prevalence and Impact on Cardiovascular Risk Profile
Brief Title: Comorbid Insomnia and Sleep Disordered Breathing in Patients Undergoing Cardiac Rehabilitation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Sleep Number, Inc. (Unknown)
Responsible Party: Principal Investigator, Amanda R. Bonikowske, Assistant Professor of Medicine, Mayo Clinic
Other Study IDs: 21-002556
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease; Sleep Disorder; Breathing-Related; Sleep Disorder; Insomnia Type
MeSH Terms: conditions — Coronary Artery Disease; Sleep Wake Disorders | interventions — Actigraphy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — about 7 tablespoons of fasting blood drawn
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polysomnograpy — Home polysomnography will be conducted using the scalable, modular Embletta system. Trained staff will instrument the participants in the evening and perform biocalibration to ensure optimal data quality
Diagnostic Test: actigraphy — A water resistant accelerometer with light sensor and event marker will be worn on the nondominant wrist for approximately 7 days. Activity counts from the device will be analyzed by proprietary software algorithms for determination of the following: sleep onset, sleep offset, total sleep time, total wake time, and sleep efficiency.16 Daytime sleep periods will be also scored to determine frequency and duration of naps. Daily data will be averaged across the 7-day period, as well as separately for weekdays and weekend, to compute measures of habitual sleep patterns.

SUMMARY:
The purpose of this research is to determine how frequently sleep disorders such as sleep disordered breathing and insomnia occur in patients with coronary artery disease enrolled in cardiac rehabilitation. By reviewing results of a variety of tests, we also hope to learn more about the cardiovascular effects on people who may have these conditions.

DETAILED DESCRIPTION:
Patients referred to the Mayo Clinic Rochester CR and meeting eligibility criteria (see Subjects section below) will be recruited and consented. Prior to beginning CR, enrolled patients will undergo baseline sleep and CV assessment at the Clinical Research and Trials Unit (CRTU). Home-based sleep monitoring will take place. Patients will also complete additional cardiometabolic and behavioral evaluation as part of the standard CR clinical care. Following completion of the 12-week CR program, a post-CR assessment may be conducted, including the same set of tests/procedures. All patients will be followed up for at least 6-months following enrollment to monitor cardiac recurrence, hospitalization and death.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be >18 years old
* Referred to CR following admitted to the hospital with a documented diagnosis of acute coronary syndrome
* Referred to CR following admission to the hospital with a documented diagnosis of ST- elevation myocardial infarction (STEMI),
* Referred to CR following admission to the hospital with a documented diagnosis of non- STEMI
* Referred to CR following admission to the hospital with a documented diagnosis of unstable angina
* Referred to CR following admission to the hospital with a documented diagnosis of post coronary artery bypass surgery
* Referred to CR following admission to the hospital after percutaneous coronary intervention (with or without stent placement).

Exclusion Criteria:

* heart failure with reduced ejection fraction
* peripheral artery disease
* valve or pericardial surgery
* heart transplantation
* patients unable to provide informed consent
* patients unable to speak and read English
* night shift workers
* pregnant women
* those who will only attend full home-based CR.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: coronary artery disease patients participating in cardiac rehab
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
To examine the prevalence of comorbid sleep disordered breathing and insomnia in post-MI patients enrolled in cardiac rehab. | 6 months
  Comorbid SDB and insomnia will be highly prevalent (>30%) in this population. Measured by home, overnight polysomnography
The combination of both sleep disorders will be associated with more detrimental CV risk markers (cardiorespiratory fitness) than either sleep disorder alone. | 6 months
  To assess whether post-MI CR patients with comorbid SDB and insomnia exhibit a more unfavorable CV profile than those without.
The combination of both sleep disorders will be associated with more detrimental CV risk markers (blood pressure) than either sleep disorder alone | 6 months
  To assess whether post-MI CR patients with comorbid SDB and insomnia exhibit a more unfavorable CV profile than those without.
The combination of both sleep disorders will be associated with more detrimental CV risk markers (lipids) than either sleep disorder alone | 6 months
  To assess whether post-MI CR patients with comorbid SDB and insomnia exhibit a more unfavorable CV profile than those without.
The combination of both sleep disorders will be associated with more detrimental CV risk markers (depression) than either sleep disorder alone | 6 months
  To assess whether post-MI CR patients with comorbid SDB and insomnia exhibit a more unfavorable CV profile than those without using the PHQ-9.
The combination of both sleep disorders will be associated with lower adherence to CR - number of attended sessions | 6 months
  To determine whether post-MI CR patients with comorbid SDB and insomnia show less adherence to CR attendance than those without
The combination of both sleep disorders will be associated with lower adherence to CR - adherence to pharmacotherapy | 6 months
  To determine whether post-MI CR patients with comorbid SDB and insomnia show less adherence to prescribed medications than those without
The combination of both sleep disorders will be associated with lower adherence to CR - exercise | 6 months
  To determine whether post-MI CR patients with comorbid SDB and insomnia show less adherence to the exercise prescription than those without
The combination of both sleep disorders will be associated with lower adherence to CR - dietary prescription | 6 months
  To determine whether post-MI CR patients with comorbid SDB and insomnia show less adherence to dietary recommendations than those without

CONTACTS AND LOCATIONS:
Overall Officials: Amanda R Bonikowske, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States